CLINICAL TRIAL: NCT07045051
Title: Effects of Fresh Mango as a Sugar Substitute Within High and Low Glycemic Breakfasts on Postprandial Glucose and Insulin
Brief Title: Glycemic/Insulinemic Effects of Fresh Mango as a Sugar Substitute in Realistic Breakfasts.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ball State University (Other)
Collaborators: National Mango Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB-FY2025-25
Record Dates: First submitted 2025-06-24; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Healthy Participants
Keywords: glycemia; insulinemia; fresh mango; vascular health
MeSH Terms: interventions — Mangifera indica extract; Dietary Sucrose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cereal Consumption with Mango (Experimental): During the Cereal and Mango arm, participants will consume a bowl of corn flakes with 2% milk sweetened with fresh mango.
  Interventions: Other: High-Glycemic Breakfast Containing Cereal and Mango
- Cereal Consumption with Table Sugar (Experimental): During the Cereal and Table Sugar arm, participants will consume a bowl of corn flakes with 2% milk sweetened with table sugar.
  Interventions: Other: High-Glycemic Breakfast Containing Cereal and Table Sugar
- Oat Consumption with Mango (Experimental): During the Oats and Mango Arm, participants will consume a bowl of oats prepared with water and sweetened with fresh mango.
  Interventions: Other: Low-Glycemic Breakfast Containing Oats and Mango
- Oat Consumption with Table Sugar (Experimental): During the Oat and Table Sugar arm, participants will consume a bowl of oats prepared with water and sweetened with table sugar.
  Interventions: Other: Low-Glycemic Breakfast Containing Oats and Table Sugar

INTERVENTIONS:
Other: Low-Glycemic Breakfast Containing Oats and Mango — Low-glycemic breakfast of 80 grams of oats prepared with 473mL water and sweetened with 146 grams of mango.
  Arms: Oat Consumption with Mango
Other: High-Glycemic Breakfast Containing Cereal and Mango — High-glycemic breakfast of 84 grams of corn flakes prepared with 355mL of 2% milk and sweetened with 262 grams of mango.
  Arms: Cereal Consumption with Mango
Other: Low-Glycemic Breakfast Containing Oats and Table Sugar — Low-glycemic breakfast of 80 grams of oats prepared with 473mL of water and sweetened with 20 grams of table sugar.
  Arms: Oat Consumption with Table Sugar
Other: High-Glycemic Breakfast Containing Cereal and Table Sugar — High-glycemic breakfast of 84 grams of corn flakes prepared with 355mL of 2% milk and sweetened with 36 grams of table sugar.
  Arms: Cereal Consumption with Table Sugar

SUMMARY:
Large blood sugar and insulin increases after meals high in table sugar are related to risk for diabetes and heart disease. Additionally, large increases in blood sugar may also negatively impact vascular health. Previous research suggests that mango consumed in small quantities has blood sugar-lowering properties, but the evidence of this within larger, more realistic meals is limited. The investigators want to understand if replacing table sugar (sucrose) with sugar from fresh mango (which also contains fiber and plant bioactives) will lead to more favorable blood sugar, insulin, and vascular responses after eating breakfast meals. The investigators will compare the postprandial glycemic, insulinemic, and vascular response to low and high glycemic meals sweetened with either fresh mango or sucrose.

DETAILED DESCRIPTION:
The investigators will recruit individuals with a BMI in the 18.5-35.0 kg/m2 range from the Ball State University campus and surrounding communities. Each participant will complete four meal trials in a randomized crossover design. At each meal trial, an intravenous catheter will be inserted and baseline blood sample collected. Brachial artery dilation will be measured using prior to the meal. Next, participants will consume one of four breakfast meals in a randomized crossover design: (1) cornflakes with 2% milk + fresh mango, (2) cornflakes with 2% milk + sucrose, (3) steel cut oats with water + fresh mango, and (4) steel cut oats with water + sucrose. Corn flakes based meals and oats based meals reflect high and low glycemic breakfasts, respectively. Within high and low glycemic meal conditions, total sugar from mango and sugar are matched, total energy is nearly identical (within 4 kcal), and macronutrients are matched.

After each meal, blood samples will be collected at the .5-, 1-, 2-, and 3-hour mark and brachial artery dilation (using the flow-mediated dilation technique) will be measured at 1-, 2-, and 3-hour marks. An acceptability survey (9-point hedonic scale) will be completed following the meal, and a satiety survey (the SLIM) will be filled out at baseline and .5-, 1-, 1.5-, 2-, 2.5-, and 3-hour mark. The investigators will measure metabolic markers (i.e., glucose, triglycerides, HDL-C) immediately after each sample collection using the Piccolo Xpress clinical chemical analyzer. Additional blood will be collected and stored as serum in order to measure insulin using commercially available ELISAs. Participants will complete a one-time DXA scan to measure body composition and bone density.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 45 years.
* Body mass index between 18.5-35.0 kg/m2
* Not pregnant (females only)
* Not postmenopausal (females only).
* Not been diagnosed with cardiovascular disease.
* Not been diagnosed with a cardiometabolic conditions (e.g., type 2 diabetes)
* Not been diagnosed with a chronic inflammatory condition (e.g., rheumatoid arthritis, inflammatory bowel disease).
* Does not regularly take anti-inflammatory drugs (more than 2x week).
* Does not use glucose-lowering drugs (e.g., metformin)
* Does not use lipid-lowering drugs (e.g., statins)
* Does not use tobacco products or any illicit drugs.
* Does not have a pacemaker.
* Can consume mango, wheat, gluten, and milk.
* Can stay in a supine position in the dark for at least ten minutes.

Exclusion Criteria:

* Not between the ages of 18-45
* Body mass index < 18.5 kg/m2 or >35.0 kg/m2
* Pregnant (females only)
* Postmenopausal status (females only).
* Been diagnosed with cardiovascular disease.
* Been diagnosed with a cardiometabolic conditions (e.g., type 2 diabetes)
* Been diagnosed with a chronic inflammatory condition (e.g., rheumatoid arthritis, inflammatory bowel disease).
* Regularly take anti-inflammatory drugs (more than 2x week).
* Uses glucose-lowering drugs (e.g., metformin)
* Uses lipid-lowering drugs (e.g., statins)
* Uses tobacco products or any illicit drugs.
* Have a pacemaker.
* Allergic to mango, wheat, gluten, and/or milk.
* Unable to lay in supine position in the dark for at least ten minutes.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Glucose | Through study completion, up to 1.5 years.
  The investigators will measure glucose at baseline and .5-, 1-, 2-, and 3-hours after each meal. These measurements will take place immediately and a complete dataset will be compiled upon study completion.
Insulin | Through study completion, up to 1.5 years.
  The investigators will measure insulin at baseline and .5- 1-, 2-, and 3-hours after each meal containing. These measurements will take place immediately and a complete dataset will be compiled upon study completion.
Flow-mediated Dilation | Through study completion, up to 1 year.
  The investigators will measure FMD at baseline and 1-, 2-, and 3-hours after the meal. These measurements will take place immediately and a complete dataset will be compiled upon study completion.

SECONDARY OUTCOMES:
HDL-C | Through study completion, up to 1 year.
  The investigators will measure HDL-C at baseline and .5-, 1-, 2-, and 3-hours after each meal. These measurements will take place immediately and a complete dataset will be compiled upon study completion.
Triglycerides | Through study completion, up to 1 year.
  The investigators will measure triglycerides at baseline and .5-, 1-, 2-, and 3-hours after each meal. These measurements will take place immediately and a complete dataset will be compiled upon study completion.
Acceptability | Through study completion, up to 1 year.
  The investigators will measure acceptability of each meal with a survey at each study visit once post-meal.
Satiety | Through study completion, up to 1 year.
  The investigators will measure satiety through a survey at baseline and at .5-, 1-, 1.5-, 2-, 2.5-, and 3-hours after the meal.

OTHER OUTCOMES:
Body Composition | Through study completion, up to 1 year.
  The investigators will measure body composition using bioelectrical impedance (InBody).
Systolic and Diastolic Pressure | Through study completion, up to 1 year.
  The investigators will measure blood pressure using an automated cuff (Omron).

CONTACTS AND LOCATIONS:
Overall Officials: Bryant Keirns, PhD, Principal Investigator — Ball State University
Locations (1):
- Health Professions Building, Ball State University, Muncie, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided